CLINICAL TRIAL: NCT03117023
Title: The Addition of Dexmedetomidine on Postoperative Sleep for Middle-aged and Elderly Patients With Gastric Cancer: A Prospective Randomized Clinical Trial
Brief Title: The Addition of Dexmedetomidine on Postoperative Sleep for Middle-aged and Elderly Patients With Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Attending, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017NLY002
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Gastric Cancer
Keywords: dexmedetomidine; sleep deprivation; gastric cancer; middle-aged and elderly patient
MeSH Terms: conditions — Stomach Neoplasms; Sleep Deprivation | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Experimental): sufentanil + dexmedetomidine
  Interventions: Drug: dexmedetomidine
- control group (No Intervention): sufentanil + saline

INTERVENTIONS:
Drug: dexmedetomidine — sufentanil 0.05ug/kh/h + dexmedetomidine 0.1ug/kg/h for 48h after surgery
  Arms: dexmedetomidine group

SUMMARY:
The purpose of this study is to find out the effect of Dexmedetomidine for treatment of sleep deprivation, pain relief and postoperative recovery on middle-aged and elderly Patients with Gastric Cancer.

DETAILED DESCRIPTION:
Patients were randomized to receive sufentanil 0.05ug/kh/h + dexmedetomidine 0.1ug/kg/h (DEX group) or sufentanil 0.05ug/kg/h + saline (control group) for 48h. The primary outcome was the total sleep time during the first three days after surgery. The secondary outcomes included pain score, daily sufentanil consumption, time to functional recovery, length of hospital stay and side effects.

ELIGIBILITY:
Inclusion Criteria:

Elective gastric cancer operation Age ≧ 55 years ASA classification：I to III, BMI: 18-30 kg/m2 without the history of gastrointestinal surgery the normal coagulation function -

Exclusion Criteria:

the history of gastrointestinal surgery Gastrostomy and jejunostomy sleep apnea syndrome or severe osahs Severe liver and heart dysfunction Severe mental illness

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2017-05-15 (Estimated); Study Completion 2017-06-01 (Estimated)

PRIMARY OUTCOMES:
sleep time | during the first three days after surgery
  total sleep time during the first three days after surgery

SECONDARY OUTCOMES:
pain score | during the first three days after surgery
  pain score measure
daily sufentanil consumption | during the first three days after surgery
  daily sufentanil consumption
functional recovery | during the first three days after surgery
  time to functional recovery
length of hospital stay | during the first three days after surgery
  length of hospital stay
side effects | during the first three days after surgery
  lethargy and mental sluggishness